CLINICAL TRIAL: NCT00548756
Title: A Phase III Prospective Randomized Trial Comparing Radiosurgery With Versus Without Whole Brain Radiotherapy for 1-3 Newly Diagnosed Brain Metastases
Brief Title: Randomized Trial Comparing Radiosurgery With vs Without Whole Brain Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID00-377; NCI-2012-01590 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Brain Cancer
Keywords: Brain Cancer; Whole Brain Radiation Therapy; Quality of Life; QOL; Questionnaire; Survey; WBRT
MeSH Terms: conditions — Brain Neoplasms | interventions — Observation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Brain Radiation Therapy (Experimental): Whole Brain Radiation Therapy
  Interventions: Procedure: Whole Brain Radiation Therapy; Behavioral: Questionnaire
- Observation (Other): Observation
  Interventions: Other: Observation; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Whole Brain Radiation Therapy — Whole Brain Radiation Therapy. Total dose = 30 Gy over 12 fractions at 2.5Gy per fraction.
  Other Names: WBRT
  Arms: Whole Brain Radiation Therapy
Other: Observation — Patients who did not receive whole brain radiation and develop recurrent disease shall receive treatment based on the number of lesions.
  Arms: Observation
Behavioral: Questionnaire — Questionnaire taking 40 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if your thinking ability (cognitive function) will be better preserved by delivering whole brain radiation therapy immediately after radiosurgical treatment of 1-3 brain metastases or to carefully observe patients after radiosurgery and hold back whole brain radiation therapy until the disease comes back.

DETAILED DESCRIPTION:
Before treatment starts, patients will have a complete history (including details of previous chemotherapy, radiotherapy, and surgery for systemic disease). Patients will have a complete neuropsychological exam and will have their Karnofsky Performance Score (KPS) figured out. Seven cognitive function tests and a quality of life (QOL) questionnaire will be given to the patients as well. It will take about 40 minutes to complete the QOL questionnaire.

Patients in this study will be randomly picked (as in the toss of a coin) to be in one of two treatment groups. Patients in one group will receive immediate whole brain radiation therapy. Patients in the other group will hold off on radiation and just be closely observed. There is an equal chance of being in either group.

All patients will receive radiosurgery treatment to the known metastases (1-3 lesions) at the beginning. All participants will be followed with serial diagnostic and functional MRI. Experimental functional imaging will be used to evaluate short-term memory and picture recognition as well as blood flow within the brain.

Formal neuropsychological testing will also be performed at each follow-up interval. Patients must come back at 4 months for neuropsychological testing. Patients will be seen for follow-up with neuropsychological evaluation, as well as diagnostic/function MRI at 1 , 2 , 4 , 6 , 9 , 12 , 15 , and 18 months and then every six months from then on. Each visit will require about 40 minutes of time.

Cost information related to protocol treatment and subsequent therapies will be tracked and collected for cost analysis between the two treatment groups.

Patients who did not receive whole brain radiation and develop recurrent disease shall receive treatment based on the number of lesions. If there are greater than 2 lesions, whole brain radiation will be given. If there are 1-2 lesions, patients will be randomly assigned to a local treatment (surgery or radiosurgery) or whole brain radiation therapy. Further recurrences in patients having not yet received whole brain radiation will be given this treatment at the time of recurrence.

The expected length of the study is 3.8 years with 6 months follow-up following the end of the study. Thus, the length of participation can range from 6 months for patients enrolling at the end of the study to over 4 years for patients enrolling at the beginning.

This is an investigational study. A total of 152 patients will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1)age 18 and older at time of registration. 2) recursive partitioning class (RPA) I or II. 3) 1 to 3 newly diagnosed brain metastases 4) must be eligible to have all lesions treated by SRS as determined by the radiation oncologist on the basis of location and size. 5)MRI with contrast must be performed with 1 month of registration. 6)Signed informed consent form approved by the IRB agreeing to randomization .

Exclusion Criteria:

1) prior WBRT 2) prior resection of brain metastasis, SRS or Gamma knife. 3) > 3 brain metastases present on MRI 4) lymphoma, small cell lung cancer, leukemia, germ cell tumors. 5) leptomeningeal disease. 6) unknown primary.7) RPA Class III (i.e. KPS < 70) 8) pregnancy.

Post-entry exclusion: No post-entry exclusions will be allowed after registration has occurred. All randomized patients will be included in the analysis and those lost to follow-up will be assigned the least favorable outcome (recurrence, death).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2001-01-02 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Cognitive Decline | 4 months
  Cognitive decline objectively measured by significant deterioration in HVLT-R LEARN at 4 months (i.e., a drop by at least 5 points compared to baseline). Difference between pretreatment baseline score and follow-up assessment scores determined by using the reliable change index (RCI).

CONTACTS AND LOCATIONS:
Overall Officials: David L. Grosshans, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chang EL, Wefel JS, Hess KR, Allen PK, Lang FF, Kornguth DG, Arbuckle RB, Swint JM, Shiu AS, Maor MH, Meyers CA. Neurocognition in patients with brain metastases treated with radiosurgery or radiosurgery plus whole-brain irradiation: a randomised controlled trial. Lancet Oncol. 2009 Nov;10(11):1037-44. doi: 10.1016/S1470-2045(09)70263-3. Epub 2009 Oct 2. PMID 19801201
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org